CLINICAL TRIAL: NCT02330458
Title: The Role of Small Bowel Ultrasound After Ileocolic Resection or When Starting Infliximab in Crohn's Disease Patients
Brief Title: The Role of Small Bowel Ultrasound in Initiation of Infliximab in Crohn's Disease Patients
Status: Unknown | Type: Observational
Last Known Status: Active, not recruiting
Sponsor: Cedars-Sinai Medical Center (Other)
Responsible Party: Principal Investigator, Namita Singh, M.D., Attending physician, Cedars-Sinai Medical Center
Other Study IDs: Pro00027597
Record Dates: First submitted 2014-12-31; First posted 2015-01-05 (Estimated); Last update posted 2017-07-19 (Actual); Status verified 2017-07

CONDITIONS: Inflammatory Bowel Disease; Crohn's Disease
Keywords: Inflammatory Bowel Disease; Crohn's disease; Pediatric IBD; small bowel ultrasound; infliximab
MeSH Terms: conditions — Inflammatory Bowel Diseases; Crohn Disease

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

INTERVENTIONS:
Procedure: Small bowel ultrasound — Small Bowel Ultrasound will be performed by a single radiologist using an Acuson S2000 machine with 6 MHz convex and 9 MHz linear array transducers (Siemens, Germany). Participants will be asked to not eat for at least 8 hours prior to the ultrasound, and to drink 500ml of a fluid of their choice just prior to the SBUS, for bowel distension and better visualization. Bowel wall thickness (BWT), the length of any segment of thickened bowel wall >3mm, hyperemia using doppler, and the presence of free fluid, stricture, intestinal dilation, or enlarged lymph nodes will be documented

SUMMARY:
Goal is to prospectively determine if stool calprotectin and change in bowel wall thickness and hyperemia, as seen on small bowel ultrasound, at week 0, 14, and 54 can be used to predict response at week 54 to infliximab in pediatric patients with small bowel Crohn's Disease.

DETAILED DESCRIPTION:
We will examine whether non-invasive disease monitoring tools such as bowel wall thickness as measured by small bowel ultrasound (SBUS) and mucosal inflammation as measured by fecal calprotectin, are independently associated with infliximab durability.

ELIGIBILITY:
Inclusion Criteria:

* Age 6-23 years
* Initiating Infliximab therapy
* Crohns disease involving the distal small bowel +/- proximal colon
* Willingness to undergo SBUS and fecal calprotectin collection prior to starting infliximab and again at week 14 and week 54
* Able to give consent by patient and/or legal guardian

Exclusion Criteria:

* Ulcerative colitis or non-Crohn's Disease patients
* Lack of small bowel disease
* Patients started on alternative therapy
* Unable or unwilling to provide consent

Ages: 6 Years to 23 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Study Population: Patients with Crohn's disease involving the small bowel, initiating Infliximab treatment.
Sampling Method: Non-Probability Sample
Enrollment: 20 (Estimated)
Dates: Start 2014-07 (Actual); Primary Completion 2017-05 (Actual); Study Completion 2018-05 (Estimated)

PRIMARY OUTCOMES:
Change in bowel wall thickness on small bowel ultrasound (SBUS) | 1 year
  Change in bowel wall thickness as measured on small bowel ultrasound from ultrasound performed on week 0 to ultrasound performed at week 54. Small Bowel Ultrasound will be performed by a single radiologist using an Acuson S2000 machine with 6 MHz convex and 9 MHz linear array transducers (Siemens, Germany). Participants will be asked to not eat for at least 8 hours prior to the ultrasound, and to drink 500ml of a fluid of their choice just prior to the SBUS, for bowel distension and better visualization. Bowel wall thickness (BWT), the length of any segment of thickened bowel wall >3mm, hyperemia using doppler, and the presence of free fluid, stricture, intestinal dilation, or enlarged lymph nodes will be documented.
  Univariate analyses will be performed to determine the association between bowel wall thickness on SBUS, and delta BWT (change in bowel wall thickness week 0 to week 14) and presence of remission at week 54

SECONDARY OUTCOMES:
Change in stool calprotectin | 1 year
  Change in level of stool calprotectin (lab) between week 0 and week 54. Stool will be collected within 24 hours of infusion and performed at our outpatient lab and analyzed by ELISA.
  Univariate analyses will be performed to determine the association between calprotectin level, delta calprotectin level (change in calprotectin level week 0 to week 14) and presence of remission at week 54.

CONTACTS AND LOCATIONS:
Overall Officials: Namita Singh, MD, Principal Investigator — Cedars-Sinai Medical Center
Locations (1):
- Cedars-Sinai Medical Center, Los Angeles, California, United States

REFERENCES:
- [Background] Moscandrew ME, Loftus EV Jr. Diagnostic advances in inflammatory bowel disease (imaging and laboratory). Curr Gastroenterol Rep. 2009 Dec;11(6):488-95. doi: 10.1007/s11894-009-0074-7. PMID 19903425
- [Background] Strobel D, Goertz RS, Bernatik T. Diagnostics in inflammatory bowel disease: ultrasound. World J Gastroenterol. 2011 Jul 21;17(27):3192-7. doi: 10.3748/wjg.v17.i27.3192. PMID 21912467
- [Background] Allen PB, De Cruz P, Lee WK, Taylor S, Desmond PV, Kamm MA. Noninvasive imaging of the small bowel in Crohn's disease: the final frontier. Inflamm Bowel Dis. 2011 Sep;17(9):1987-99. doi: 10.1002/ibd.21598. Epub 2011 Feb 1. PMID 21287661
- [Background] Fraquelli M, Colli A, Casazza G, Paggi S, Colucci A, Massironi S, Duca P, Conte D. Role of US in detection of Crohn disease: meta-analysis. Radiology. 2005 Jul;236(1):95-101. doi: 10.1148/radiol.2361040799. PMID 15987966
- [Background] Parente F, Molteni M, Marino B, Colli A, Ardizzone S, Greco S, Sampietro G, Foschi D, Gallus S. Are colonoscopy and bowel ultrasound useful for assessing response to short-term therapy and predicting disease outcome of moderate-to-severe forms of ulcerative colitis?: a prospective study. Am J Gastroenterol. 2010 May;105(5):1150-7. doi: 10.1038/ajg.2009.672. Epub 2009 Dec 8. PMID 19997096